CLINICAL TRIAL: NCT04734873
Title: Phase 3, Randomized, Placebo Controlled, Double-blind, Multicenter, Stratified Study of CPI-006 Plus Standard of Care Versus Placebo Plus Standard of Care in Mild to Moderately Symptomatic Hospitalized Covid-19 Patients
Brief Title: CPI-006 Plus Standard of Care Versus Placebo Plus Standard of Care in Mild to Moderately Symptomatic Hospitalized Covid-19 Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision. Not related to safety issues.
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-006-003
Record Dates: First submitted 2021-01-29; First posted 2021-02-02 (Actual); Results first posted 2022-08-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Covid-19
Keywords: SARS-CoV-2; Covid; Coronavirus; Covid19; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — CPI-006

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CPI-006 (2 mg/kg) Plus Standard of Care (Experimental): Participants will receive a single dose of CPI-006 at 2 mg/kg up to a maximum dose of 200 mg intravenously on Day 1 plus standard of care.
  Interventions: Drug: CPI-006 2 mg/kg + SOC
- CPI-006 (1 mg/kg) Plus Standard of Care (Experimental): Participants will receive a single dose of CPI-006 at 1 mg/kg up to a maximum dose of 100 mg intravenously on Day 1 plus standard of care.
  Interventions: Drug: CPI-006 1 mg/kg + SOC
- Placebo Plus Standard of Care (Placebo Comparator): Participants will receive a single dose of placebo intravenously on Day 1 plus standard of care.
  Interventions: Drug: Placebo + SOC

INTERVENTIONS:
Drug: CPI-006 2 mg/kg + SOC — IV CPI-006 2 mg/kg up to a maximum dose of 200 mg plus standard of care
  Arms: CPI-006 (2 mg/kg) Plus Standard of Care
Drug: CPI-006 1 mg/kg + SOC — IV CPI-006 1 mg/kg up to a maximum dose of 100 mg plus standard of care
  Arms: CPI-006 (1 mg/kg) Plus Standard of Care
Drug: Placebo + SOC — IV placebo plus standard of care
  Arms: Placebo Plus Standard of Care

SUMMARY:
This is a phase 3, randomized, placebo controlled, double-blind, multicenter, stratified study of CPI-006 plus standard of care (SOC) versus placebo plus SOC in mild to moderately symptomatic hospitalized Covid-19 patients with the primary objective to compare the proportion of participants alive and respiratory failure free between CPI-006 plus SOC versus placebo plus SOC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed positive by polymerase chain reaction (PCR) or antigen test for SARS-CoV-2 with sample collection ≤ 10 days prior to randomization
* Covid-19 illness of any duration of symptoms
* Hospitalized for Covid-19 for ≤ 5 days with mild to moderate Covid-19 symptoms and meets criteria for either Category 4, Category 5, or Category 6 per 8-point ordinal scale
* Adequate organ function
* Participants of child-bearing age must agree to use adequate contraception for 6 weeks after study treatment administration

Exclusion Criteria:

* Signs of acute respiratory distress syndrome or respiratory failure necessitating mechanical ventilation at time of screening/randomization or anticipated need for mechanical ventilation
* History of severe chronic respiratory disease and requirement for long-term oxygen therapy
* Uncontrolled active systemic infection or hemodynamic instability requiring admission to an intensive care unit
* Malignant tumor receiving treatment, or other serious systemic diseases affecting life expectancy within 29 days of screening
* Receipt of cancer chemotherapy or immunomodulatory drugs during preceding 2 months (steroids for treatment of Covid-19 are acceptable)
* Convalescent plasma (CCP) or anti-SARS-CoV-2 monoclonal antibodies administered <24 hours prior to randomization. Must have recovered from any adverse events related to CCP treatment. Received chloroquine or hydroxychloroquine within last 7 days or during the study
* Current participation in other clinical trials including extended access programs
* Active deep vein thrombosis or pulmonary embolism within last 6 months
* Anticipated discharge from hospital or transfer to another hospital which is not a study site within 48 hours of admission
* Active uncontrolled co-morbid disease that may interfere with study conduct or interpretation of findings
* Known to be positive for HIV or positive test for chronic HBV infection or positive test for hepatitis C antibody
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Mahabhashyam, MD, MPH, Study Chair — Corvus Pharmaceuticals
Locations (91):
- United States (13):
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - El Centro Regional Medical Center, El Centro, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Torrance Memorial Medical Center, Torrance, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cambridge Medical Trials, Alexandria, Louisiana
  - MedPharmics, Metairie, Louisiana
  - Holy Cross Hospital, Silver Spring, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Stony Brook University Medical Center, Stony Brook, New York
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
- Argentina (13):
  - Clinica Zabala, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clínica Adventista Belgrano, Estomba, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Clinica Independencia, Munro, Buenos Aires
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Centro de Investigación Clínica - Clínica Viedma, Viedma, Río Negro Province
  - Centro Médico IPAM, Rosario, Santa Fe Province
  - Hospital Provincial Del Centenario, Rosario, Santa Fe Province
  - Clinica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - Hospital de Clínicas Presidente Dr. Nicolás Avellaneda, San Miguel de Tucumán, Tucumán Province
  - Fundación Sanatorio Güemes, Buenos Aires
  - Sanatorio Finochietto, Buenos Aires
  - Hospital Rawson, Córdoba
- Brazil (12):
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Hospital Agamenon Magalhães, Recife, Pernambuco
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão, Blumenau, Santa Catarina
  - Clínica Supera, Chapecó, Santa Catarina
  - Centro Hospitalar Nossa Saúde, Curitiba
  - Universidade Municipal São Caetano do Sul, São Caetano do Sul
  - Conjunto Hospitalar do Mandaqui, São Paulo
  - Hospital Anchieta, São Paulo
  - Hospital de Base Da Faculdade de Medicina de São José Do Rio Preto, São Paulo
  - Hospital E Maternidade Celso Pierro PUCCAMP, São Paulo
  - Universidade Federal Do Espirito Santo - Hospital Universitário Cassiano Antônio de Moraes - HUCAM, Vitória
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- Chile (4):
  - Hospital Base de Osorno, Concepción
  - Clinica Vespucio, La Florida
  - Research Network Consulting, Linares
  - Clínica Dávila Y Servicios Médicos SA, Santiago
- Colombia (9):
  - Rodrigo Botero S.A.S, Medellín, Antioquia
  - Fundacion Santa Fe de Bogota, Bogotá, Cundinamarca
  - Clínica Universidad De la Sabana, Chía, Cundinamarca
  - Fundacion Centro de Excelencia en Enfermedades Cronicas No Transmisibles, Montería, Departamento de Córdoba
  - Clínica de la Mujer S.A.S., Bogotá
  - Hospital Universitario Clinica San Rafael, Bogotá
  - Fundacion Hospitalaria San Vicente de Paul, Medellín
  - Promotora Medica Las Américas S.A- Clínica Las Américas, Medellín
  - Fundación Valle Del Lili, Santiago de Cali
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany
- Italy (8):
  - Azienda Ospedaliera Cotugno, Napoli, Campania
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan, Lombardy
  - ASST Santi Paolo e Carlo - Azienda Universitaria-Polo Universitario San Paolo, Milan, Lombardy
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - ASST della Valle Olona - Azienda Ospedaliera Ospedale Di Circolo Di Busto Arsizio, Busto Arsizio
- Mexico (4):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey, Nuevo León
  - Hospital Civil de Culiacán, Culiacán, Sinaloa
  - Hospital General de Culiacán, Culiacán, Sinaloa
- Peru (10):
  - Hospital Nacional Sergio E. Bernales, Comas, Lima region
  - Hospital Chancay y Servicios Basicos de Salud, Huaral, Lima region
  - Hospital Central Fuerza Aérea del Perú, Miraflores, Lima region
  - Hospital María Auxiliadora, San Juan de Miraflores, Lima region
  - Clínica Providencia, San Miguel, Lima region
  - Clínica San Pablo, Santiago de Surco, Lima region
  - Hospital Alberto Sabogal Sologuren, Callao
  - Hospital Nacional Adolfo Guevara Velasco Essalud, Cusco
  - Hospital Militar Central, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Spain (6):
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Universitario A Coruña, Santiago de Compostela
- Ukraine (9):
  - Municipal Institution City Clinical Hospital #6 of Dnipropetrovsk Regional Council, Dnipro, Dnipropetrovsk Oblast
  - Kharkiv Regional Clinical Infectious Diseases Hospital, Kharkiv, Kharkivs’ka Oblast’
  - Poltava Regional Clinical Infectious Hospital, Poltava, Poltava Oblast
  - Communal Non-Commercial Enterprise Vinnytsia City Clinical Hospital 1, Vinnytsia, Vinnytsia Oblast
  - Municipal enterprise Volyn Regional Clinical Hospital of Volyn Regional Council, Lutsk, Volyn Oblast
  - MNPE City Hospital No. 6 of Zaporizhzhia City Council, Zaporizhzhia, Zaporizhzhia Oblast
  - Municipal Institution City Hospital #7, Zhaporizhzhya, Zaporizhzhia Oblast
  - CNPE City Clinical Hospital #3 of Chernivtsi City Council, Chernivtsi
  - Municipal Non-profit Enterprise "City Clinical Hospital # 4" of Dnipro City Council, Dnipro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 participants were screened and 42 were randomized. Of the 42 participants randomized, only 40 received the treatment assigned at randomization (2 were randomized but withdrew consent prior to receiving study treatment).
Groups:
- Treatment A: CPI-006 2 mg/kg + SOC: IV CPI-006 2 mg/kg up to a maximum dose of 200 mg on Day 1 plus standard of care
- Treatment B: CPI-006 1 mg/kg + SOC: IV CPI-006 1 mg/kg up to a maximum dose of 100 mg on Day 1 plus standard of care
- Treatment C: Placebo + SOC: IV placebo on Day 1 plus standard of care
Period: Overall Study
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC
Started | 16 | 14 | 12
Completed | 14 | 11 | 9
Not Completed | 2 | 3 | 3
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Randomized but not dosed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 42 participants were randomized however only 40 received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC | Total
Number analyzed (Participants) | 16 | 14 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 12 | 38
  >=65 years | 3 | 1 | 0 | 4
Age, Continuous [Median (Full Range); unit: years] | 56.5 [28 to 69] | 53.0 [25 to 67] | 55.0 [21 to 63] | 56.0 [21 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9 | 18
  Male | 10 | 11 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 3 | 12
  Not Hispanic or Latino | 8 | 11 | 8 | 27
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 13 | 11 | 9 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 13 | 12 | 41
  Spain | 0 | 1 | 0 | 1
8-point Ordinal Scale Assessment [Count of Participants; unit: Participants] — Scale categories: 1=Not hospitalized, no limitations on activities; 2=Not hospitalized, limitation on activities and/or requiring home oxygen; 3=Hospitalized, not requiring supplemental oxygen - no longer requiring ongoing medical care; 4=Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (Covid-19 related or otherwise); 5=Hospitalized, requiring supplemental oxygen; 6=Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7=Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation; 8=Death
  Participants
    4 | 0 | 3 | 2 | 5
    5 | 7 | 10 | 7 | 24
    6 | 9 | 1 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Alive and Respiratory Failure Free of CPI-006 Plus SOC Versus Placebo Plus SOC
Description: Proportion of participants who are alive and free from respiratory deterioration in each active arm compared to placebo arm as measured by the modified World Health Organization (WHO) 8-point Ordinal Scale for Clinical Improvement in which: 1=Not hospitalized, no limitations on activities; 2=Not hospitalized, limitation on activities and/or requiring home oxygen; 3=Hospitalized, not requiring supplemental oxygen - no longer requiring ongoing medical care; 4=Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (Covid-19 related or otherwise); 5=Hospitalized, requiring supplemental oxygen; 6=Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7=Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation; 8=Death.
Time Frame: During the 28 days after dosing
Population: All participants who received any amount of study drug (CPI-006 or placebo) and have post-baseline efficacy assessment based on the 8-point ordinal scale.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC
Number analyzed (Participants) | 15 | 14 | 11
Participants | 14 | 12 | 9

2. Secondary Outcome: Time to Recovery of CPI-006 Plus SOC Versus Placebo Plus SOC
Description: Time to recovery after dosing in each active arm compared to placebo arm as measured by the modified WHO 8-point Ordinal Scale for Clinical Improvement in which: 1=Not hospitalized, no limitations on activities; 2=Not hospitalized, limitation on activities and/or requiring home oxygen; 3=Hospitalized, not requiring supplemental oxygen - no longer requiring ongoing medical care; 4=Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (Covid-19 related or otherwise); 5=Hospitalized, requiring supplemental oxygen; 6=Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7=Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation; 8=Death.
Time Frame: During the 28 days after dosing
Population: All participants who received any amount of study drug (CPI-006 or placebo) and recovered during the 28 days after dosing.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC
Number analyzed (Participants) | 14 | 14 | 10
days | 6.0 [4.0 to 9.0] | 4.5 [3.0 to 8.0] | 7.0 [2.0 to 12.0]

3. Secondary Outcome: Time to Clinical Improvement of CPI-006 Plus SOC Versus Placebo Plus SOC
Description: Time to clinical improvement in each active arm compared to placebo arm as measured by the modified WHO 8-point Ordinal Scale for Clinical Improvement in which: 1=Not hospitalized, no limitations on activities; 2=Not hospitalized, limitation on activities and/or requiring home oxygen; 3=Hospitalized, not requiring supplemental oxygen - no longer requiring ongoing medical care; 4=Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (Covid-19 related or otherwise); 5=Hospitalized, requiring supplemental oxygen; 6=Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7=Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation; 8=Death. Clinical improvement is defined as ≥ 2 points improvement in the 8-point ordinal scale.
Time Frame: During the 28 days after dosing
Population: All participants who received any amount of study drug (CPI-006 or placebo) and achieved clinical improvement during the 28 days after dosing.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC
Number analyzed (Participants) | 14 | 14 | 11
days | 6.0 [4.0 to 9.0] | 4.5 [3.0 to 8.0] | 7.0 [2.0 to 12.0]

4. Secondary Outcome: Mortality Rate Due to Any Cause of CPI-006 Plus SOC Versus Placebo Plus SOC
Description: Proportion of participants who died in each active arm compared to placebo arm
Time Frame: During the 28 days after dosing
Population: All participants who received any amount of study drug (CPI-006 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC
Number analyzed (Participants) | 15 | 14 | 11
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From initiation of study treatment through study Day 28 (4 weeks)
Description: The Safety Population includes all participants who received any amount of study treatment (CPI-006, placebo, or SOC).
Arm/Group | Treatment A: CPI-006 2 mg/kg + SOC | Treatment B: CPI-006 1 mg/kg + SOC | Treatment C: Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 2/11
Other Adverse Events (participants affected / at risk) | 5/15 | 2/14 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: CPI-006 2 mg/kg + SOC (N=15) | Treatment B: CPI-006 1 mg/kg + SOC (N=14) | Treatment C: Placebo + SOC (N=11)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: CPI-006 2 mg/kg + SOC (N=15) | Treatment B: CPI-006 1 mg/kg + SOC (N=14) | Treatment C: Placebo + SOC (N=11)
Myopia (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to enrollment difficulties and, as a result, some of the originally planned efficacy analyses could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are free to publish/present study results from their site upon occurrence of one of either: a multi-center publication, no publication is submitted within 18 months after end of study, or sponsor confirms there will be no publication. Investigators must provide the sponsor all draft publications for review at least 30 days prior to submission. Sponsor may request to defer publication and/or delete sponsor's confidential information to allow the sponsor to preserve its IP rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04734873/Prot_SAP_000.pdf